CLINICAL TRIAL: NCT04246905
Title: Efficacy of Adjunctive Sulforaphane for Depression: Study Protocol for a Randomized, Double-blind, Placebo-controlled Study
Brief Title: A 12-weeks Study to Evaluate Sulforaphane in the Treatment of Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019209
Record Dates: First submitted 2020-01-06; First posted 2020-01-29 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Depressive Disorder
Keywords: Sulforaphane; Depression; Fatigue; Cognition
MeSH Terms: conditions — Depressive Disorder; Depression; Fatigue | interventions — sulforaphane; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Intervention Model Description: Patients will be treated with sulforaphane or placebo for 12 weeks after ramdomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and researchers are blind to treatment allocation (double-blind). An independent researcher developed the computer-generated randomization plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- sulforaphane (Active Comparator): sulforaphane treatment arm
  Interventions: Drug: sulforaphane; Drug: selective 5 - HT reuptake inhibitors (SSRI)
- placebo (Placebo Comparator): placebo arm
  Interventions: Other: placedo; Drug: selective 5 - HT reuptake inhibitors (SSRI)

INTERVENTIONS:
Drug: sulforaphane — To examine the add-on effect of sulforaphane in depression patients with selective 5 - HT reuptake inhibitors (SSRI) treatment
  Arms: sulforaphane
Other: placedo — To examine the add-on effect of sulforaphane in depression patients with selective 5 - HT reuptake inhibitors (SSRI) treatment
  Arms: placebo
Drug: selective 5 - HT reuptake inhibitors (SSRI) — To examine the add-on effect of sulforaphane in depression patients with selective 5 - HT reuptake inhibitors (SSRI) treatment

SUMMARY:
Major depressive disorder is a serious, recurrent and disabling mental disorder, which is the second leading cause of years lost to disability worldwide. Accumulating evidence suggests the important role for inflammation and oxidative stress in the pathophysiology of depression. Sulforaphane extracted from broccoli sprout is an agent with potent anti-oxidant and anti-inflammatory activity. Previous studies suggested sulforaphane activates Keap1-Nrf2 system to prevent depression-like phenotype in mice. In this study, the investigator attempts to evaluate the efficacy, safety, and tolerability of sulforaphane plus a fixed oral antipressant in adult participants diagnosed with depression.

DETAILED DESCRIPTION:
A total of 90 patients aged 18-55 years with depression will be included, all of whom gave informed consent. Participants will receive 12 weeks of either sulforaphane or placebo per day, in addition to the existing treatment. Baseline assessments include demographics, a comprehensive medical history, anthropometric measurements (weight and height), physical examination, and lab work. Clinical symptoms will be assessed by the Montgomery-A° sberg Depression Rating Scale (MADRS), Hamilton depressive scale (HAMD), Hamilton Anxiety Scale(HAMA), and Patient Health Questionnaire-9 (PHQ-9). The safety will be assessed by Treatment Emergent Symptom Scale (TESS). The cognitive function will be evaluated by MATRICS Consensus Cognitive Battery （MCCB）at the beginning of the study and at week 12. The cranial MRI is examined at baseline and repeated at week 12. The primary outcomes will be the effective time and the percentages of efficacy at 8 weeks, measured using the MADRS. Efficacy is defined as ≥50% decreases in the total score of MADRS. Secondary outcomes include global psychopathology, quality of life, functioning, cognition, biological data, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Clinical diagnosis of recurrent MDD or single-episode MDD with MADRS≥22, CGI-SI≥4
* be adherent to the continued oral antidepressant treatment medication

Exclusion Criteria:

* treatment-resistant depression
* have known allergies, hypersensitivity, intolerance, or contraindications to SSRI or any of the trial preparations
* strong homicidal ideation/intent
* pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Montgomery-A° sberg Depression Rating Scale (MADRS) total score at week 8 | baseline and week 8
  Range from 0-60, higher score indicates more severe symptoms

SECONDARY OUTCOMES:
Changes of Hamilton depressive scale (HAMD) from baseline to week 12 | Week 0 and week 12.
  Range from 24-75, higher score indicates more severe symptoms
the total scores of Hamilton depressive scale (HAMD) | Week 0, 2, 4, 6, 8, 12.
  Range from 24-75, higher score indicates more severe symptoms
Hamilton Anxiety Scale(HAMA) | Week 0, 2, 4, 6, 8, 12.
  Range from 0-56, higher score indicates more severe symptoms
The total score of clinical global impression-severty of illness (CGI-SI) | Week 0, 2, 4, 6, 8, 12.
  Range from 0-7, higher score indicates more severe symptoms
Change of MATRICS Consensus Cognitive Battery （MCCB）from baseline to week 12 | Week 0, 12.
  To evaluate the efficacy of adjunctive sulforaphane treatment in improving cognitive functions. Higher score indicates better cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute of Second Xiangya Hospital,CSU, Changsha, Hunan, China